CLINICAL TRIAL: NCT06073288
Title: Unveiling the Microbial Impact on Intestinal Fibrosis: New Insights for the Pathogenesis and Treatment of Crohn's Disease-associated Complications
Brief Title: Unveiling the Microbial Impact on Intestinal Fibrosis
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Silvio Danese, Director of Gastroenterology and Endoscopy Unit, IRCCS San Raffaele
Other Study IDs: RF-2021-12372637
Record Dates: First submitted 2023-09-25; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Crohn's Disease (CD): 15 CD patients (5 patients/stage: (B1 (more inflammatory, non-structuring), B2 (structuring, non-penetrating) and B3 (structuring and penetrating).
  Patient stratification is based on previous classifications done in accordance with the standard of care through TC, RMI or Ecography. For this reason, patients classification is known before surgery.
  Interventions: Other: Surgical specimens of CD and no-IBD patients
- non-Intestinal Bowel Disease patients (no-IBD): 5 patients without IBD-related diseases (ex. diverticulitis)
  Interventions: Other: Surgical specimens of CD and no-IBD patients

INTERVENTIONS:
Other: Surgical specimens of CD and no-IBD patients — Specimens of CD patients and patients without IBD-related disease (ex. diverticulitis) will be collected during the surgery, without other risks for the patients, since we will use only material left after pathologist analysis

SUMMARY:
Crohn's disease (CD), belonging to the class of Inflammatory Bowel Diseases, is a chronic inflammatory disorder that may affect any location of the gastrointestinal tract. It is characterized by transmural inflammation and an overwhelming immune response of the gut mucosa, which leads to severe clinical symptoms. More than 50% of CD patients develop a penetrating or stricturing disease due to fibrostenosis, which most of the time requires surgical intervention since no therapies have been found as effective yet. Among the histological features of stricturing CD, the thickening of the muscularis mucosae and muscularis propria is the main hallmark, primarily due to the excessive proliferation of mesenchymal cells and the increased accumulation of a collagen-rich extracellular matrix in the submucosa, caused by multiple mechanisms, including i) the proliferation of existing local fibroblasts, the induction of both ii) epithelial-to-, and iii) endothelial-to-mesenchymal transition. Even if the alteration of these mucosal functions is mainly caused by the continuous tissue injury occurring during CD-associated chronic inflammation, recent reports suggested that CD associated fibrosis may be driven by inflammation-independent triggers, such as microbiota dysbiosis.

Shedding the light on this aspect of CD fibrosis may lead to the development of innovative therapeutic strategies eventually blocking the gut thickening.

DETAILED DESCRIPTION:
This is a cross-sectional observational study involving patients with Crohn's Disease (CD) (n=15) and patients with non-Intestinal Bowel Disease (IBD) (n=5) undergoing surgery in the Gastroenterology and Digestive Endoscopy unit within Gastro Center (IRCCS Ospedale San Raffaele) according to the standard of care.

Specimens will be collected during the surgery, without other risks for the patients, since we will use only material left after pathologist analysis.

CD-derived surgical specimens will be processed to obtain a cell suspension, that will be frozen and stored for the following cell sorting. For non-IBD tissue processing, each surgical specimen will be cut into two pieces. One will be processed to obtain the cell suspension to be stored, whereas the remaining tissue will be processed to isolate lamina propria fibroblasts and endothelial cells, as well as to generate epithelial organoids.

Ospedale San Raffaele (OSR - Operative Unit (UO)1 (UO1)) is the promoter of this study. The other center participating in the study is University of Milan (UO2), which has in charge the development of 3D microfluidic devices for the in vitro experiments. Patients will be enrolled only in UO1.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 and <70 years
* All patients will sign the informed consent
* Given that it is an observational study, also pregnant and breastfeed patients could be included

Additionally, for CD patients:

- classification on different stages: (B1 (more inflammatory, non-structuring), B2 (structuring, non-penetrating) and B3 (structuring and penetrating). Patient stratification is based on previous classifications done in accordance with the standard of care through TC, RMI or Ecography.

Additionally, for non-IBD patients:

- subjects undergoing surgery for non-IBD diseases (ex. diverticulitis) in accordance with the standard of care

Exclusion Criteria:

For CD patients:

* CD subjects without previously classification in B1, B2, B3
* Patients <18 years or > 70 years
* Patients without the signed informed consent

For non-IBD patients:

* Patients <18 years or > 70 years
* Patients without the signed informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients undergoing surgery:
  - 15 CD patients (5 patients/stage: (B1 (more inflammatory, non-structuring), B2 (structuring, non-penetrating) and B3 (structuring and penetrating).
  Patient stratification is based on previous classifications done in accordance with the standard of care through TC, RMI or Ecography. For this reason, patients classification is known before surgery.
  - 5 patients without IBD-related diseases (ex. diverticulitis)
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
To perform flow cytometry, RNAseq, metatranscriptomics, transcriptomics and lipidomics on CD and non-IBD cells | 1-36 months
  To evaluate how bacterial factors may impact the transcriptomic state of the different host cell compartments in terms of profibrotic pathway and gene activation. Cells will undergo FACS for CD31, EpCam, and CD90 markers for isolating endothelial cells, epithelial cells, and fibroblasts, respectively, as the well-known cellular players in the fibrotic process. Single-cell populations will undergo library preparation and will be analyzed by ribo-minus RNAseq at 30M reads of depth. Metatranscriptomics for profiling the microbial composition, as well as the transcriptomics to determine both the differential gene expression (DGE) and the Gene Set Enrichment Analysis (GSEA) will be performed. The relative abundances of Brevibacteriaceae, Caulobacteraceae, and Sphingomonadaceae-derived factors will be calculated using Kraken2 to identify which cell subtype(s) among CD-derived fibroblasts, endothelial cells, and epithelial organoids harbor(s) the fibrotic-specific microbial composition.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided